CLINICAL TRIAL: NCT05874700
Title: A Pilot Study of Perioperative Application of Sivelestat Sodium in Acute Type A Aortic Dissection Patients With Preoperative Moderate to Severe Hypoxemia to Shorten the Duration of Postoperative Invasive Mechanical Ventilation
Brief Title: A Pilot Study of Sivelestat Sodium to Shorten Mechanical Ventilation in Acute Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaotong Hou (Other)
Responsible Party: Sponsor-Investigator, Xiaotong Hou, Clinical Professor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-4
Record Dates: First submitted 2023-05-06; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Acute Aortic Dissection
Keywords: acute type A aortic dissection; preoperative moderate to severe hypoxemia; sivelestat sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sivelestat sodium group (Experimental): sivelestat sodium
  Interventions: Drug: Sivelestat sodium was given intravenously
- Placebo control group (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo was given intravenously

INTERVENTIONS:
Drug: Sivelestat sodium was given intravenously — Anesthesia induction began with a 0.2mg/Kg/h pump test drug until 48 hours after endotracheal intubation was removed or up to 7 days. If the patient was judged to have successfully removed the endotracheal tube, drug administration was discontinued; If the endotracheal intubation was not removed successfully up to 7 days, drug administration was also discontinued. During CPB, 0.1mg/100mL of the experimental drug was injected into the circulating pump immediately after CPB began.
  Other Names: Sivelestat sodium group
  Arms: Sivelestat sodium group
Drug: Placebo was given intravenously — Anesthesia induction began with a 0.2mg/Kg/h pump test drug until 48 hours after endotracheal intubation was removed or up to 7 days. If the patient was judged to have successfully removed the endotracheal tube, drug administration was discontinued; If the endotracheal intubation was not removed successfully up to 7 days, drug administration was also discontinued. During CPB, 0.1mg/100mL of the experimental drug was injected into the circulating pump immediately after CPB began.
  Other Names: Placebo control group
  Arms: Placebo control group

SUMMARY:
This is A prospective, randomized, placebo-controlled, reestimable adaptive clinical study to evaluate the efficacy and safety of perioperative application of sivelestat sodium to shorten the duration of postoperative invasive mechanical ventilation in acute type A aortic dissection patients with preoperative moderate and severe hypoxemia (PaO2/FiO2≤200mmHg).

DETAILED DESCRIPTION:
In recent years, sivelestat sodium therapy has been used to treat and prevent CPB-associated lung injury with good results. Morimoto K et al., randomized control of a small sample size, demonstrated that sivelestat sodium improves respiratory function in patients with severe respiratory failure after hypothermia thoracic aortic surgery. A retrospective study by Morimoto N et al. confirmed that prophylactic application of sivelestat sodium at the beginning of CPB could improve postoperative respiratory function and shorten the duration of mechanical ventilation in patients with hypothermic circulatory arrest. At present, there is a lack of reliable RCTS to confirm that the intraoperative application of sivelestat sodium can effectively treat preoperative acute lung injury, improve CPB-related lung injury, and reduce the incidence of postoperative acute lung injury. Therefore, the objective of this study was to design A randomized controlled study to evaluate the clinical efficacy and safety of intraoperative use of sivelestat sodium to shorten the duration of postoperative invasive mechanical ventilation in acute type A aortic dissection patients with preoperative moderate to severe hypoxemia. The purpose of this preliminary clinical trial is to provide theoretical basis for sample size calculation of randomized controlled trials, and to evaluate the scientific nature and feasibility of randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75;
2. Spontaneous acute (≤14 days) type A aortic dissection;
3. In the emergency department, hypothermic circulatory arrest combined with unilateral anterograde cerebral perfusion was expected to be performed on the aortic arch surgery;
4. Preoperative PaO2/FiO2≤200mmHg;

Exclusion Criteria:

1. Preoperative cardiogenic shock;
2. preoperative liver insufficiency;
3. Preoperative dissection involves important organs and seriously endangers the patient's life
4. Pregnant women;
5. hereditary connective tissue diseases, such as Marfan syndrome, Ehlers-Danlos syndrome, Loeys-Dietz syndrome, etc.;
6. Behcet's disease;
7. aortitis;
8. There is a history of neurologic disease that has been clearly diagnosed;
9. There is a history of a clearly diagnosed mental illness;
10. There is a definite diagnosis of chronic respiratory disease;
11. There is a clearly diagnosed immune disease;
12. There is a definite diagnosis of hematological diseases;
13. severe renal failure or require dialysis treatment;
14. Taking anti-inflammatory or anti-coagulant drugs within a week before admission;
15. People who are allergic to sivelestat sodium and other ingredients;
16. Has participated in other clinical trials;
17. The clinician judges that it is not suitable for inclusion in the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Invasive mechanical ventilation time | 28 days after surgery
  Duration from the initiation of invasive mechanical ventilation to the first successful removal of the endotracheal tube

SECONDARY OUTCOMES:
Total invasive mechanical ventilation | 28 days after surgery
  mode and duration
Total non-invasive mechanical ventilation | 28 days after surgery
  mode and duration
Total high flow oxygen uptake | 28 days after surgery
  mode and duration
Oxygenation index and area under curve | 28 days after surgery
  Oxygenation index
PaO2/FiO2≤300mmHg Duration | 28 days after surgery
  Duration of hypoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomeng Wang, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bossone E, Eagle KA. Epidemiology and management of aortic disease: aortic aneurysms and acute aortic syndromes. Nat Rev Cardiol. 2021 May;18(5):331-348. doi: 10.1038/s41569-020-00472-6. Epub 2020 Dec 22. PMID 33353985
- [Result] Guo Z, Yang Y, Zhao M, Zhang B, Lu J, Jin M, Cheng W. Preoperative hypoxemia in patients with type A acute aortic dissection: a retrospective study on incidence, related factors and clinical significance. J Thorac Dis. 2019 Dec;11(12):5390-5397. doi: 10.21037/jtd.2019.11.68. PMID 32030257
- [Result] Liu N, Zhang W, Ma W, Shang W, Zheng J, Sun L. Risk factors for hypoxemia following surgical repair of acute type A aortic dissection. Interact Cardiovasc Thorac Surg. 2017 Feb 1;24(2):251-256. doi: 10.1093/icvts/ivw272. PMID 27756811
- [Result] Wang Y, Xue S, Zhu H. Risk factors for postoperative hypoxemia in patients undergoing Stanford A aortic dissection surgery. J Cardiothorac Surg. 2013 Apr 30;8:118. doi: 10.1186/1749-8090-8-118. PMID 23631417
- [Result] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Result] Duan XZ, Xu ZY, Lu FL, Han L, Tang YF, Tang H, Liu Y. Inflammation is related to preoperative hypoxemia in patients with acute Stanford type A aortic dissection. J Thorac Dis. 2018 Mar;10(3):1628-1634. doi: 10.21037/jtd.2018.03.48. PMID 29707315
- [Result] Oda S, Aibiki M, Ikeda T, Imaizumi H, Endo S, Ochiai R, Kotani J, Shime N, Nishida O, Noguchi T, Matsuda N, Hirasawa H; Sepsis Registry Committee of The Japanese Society of Intensive Care Medicine. The Japanese guidelines for the management of sepsis. J Intensive Care. 2014 Oct 28;2(1):55. doi: 10.1186/s40560-014-0055-2. eCollection 2014. PMID 25705413
- [Result] Hashimoto S, Okayama Y, Shime N, Kimura A, Funakoshi Y, Kawabata K, Ishizaka A, Amaya F. Neutrophil elastase activity in acute lung injury and respiratory distress syndrome. Respirology. 2008 Jun;13(4):581-4. doi: 10.1111/j.1440-1843.2008.01283.x. Epub 2008 Apr 10. PMID 18410258
- [Result] Polverino E, Rosales-Mayor E, Dale GE, Dembowsky K, Torres A. The Role of Neutrophil Elastase Inhibitors in Lung Diseases. Chest. 2017 Aug;152(2):249-262. doi: 10.1016/j.chest.2017.03.056. Epub 2017 Apr 23. PMID 28442313
- [Result] Kotani M, Kotani T, Ishizaka A, Fujishima S, Koh H, Tasaka S, Sawafuji M, Ikeda E, Moriyama K, Kotake Y, Morisaki H, Aikawa N, Ohashi A, Matsushima K, Huang YC, Takeda J. Neutrophil depletion attenuates interleukin-8 production in mild-overstretch ventilated normal rabbit lung. Crit Care Med. 2004 Feb;32(2):514-9. doi: 10.1097/01.CCM.0000110677.16968.E4. PMID 14758172
- [Result] Miyoshi S, Hamada H, Ito R, Katayama H, Irifune K, Suwaki T, Nakanishi N, Kanematsu T, Dote K, Aibiki M, Okura T, Higaki J. Usefulness of a selective neutrophil elastase inhibitor, sivelestat, in acute lung injury patients with sepsis. Drug Des Devel Ther. 2013 Apr 10;7:305-16. doi: 10.2147/DDDT.S42004. Print 2013. PMID 23596346
- [Result] Morimoto K, Nishimura K, Miyasaka S, Maeta H, Taniguchi I. The effect of sivelestat sodium hydrate on severe respiratory failure after thoracic aortic surgery with deep hypothermia. Ann Thorac Cardiovasc Surg. 2011;17(4):369-75. doi: 10.5761/atcs.oa.10.01555. PMID 21881324
- [Result] Morimoto N, Morimoto K, Morimoto Y, Takahashi H, Asano M, Matsumori M, Okada K, Okita Y. Sivelestat attenuates postoperative pulmonary dysfunction after total arch replacement under deep hypothermia. Eur J Cardiothorac Surg. 2008 Oct;34(4):798-804. doi: 10.1016/j.ejcts.2008.07.010. Epub 2008 Aug 22. PMID 18722781
- [Result] Ryugo M, Sawa Y, Takano H, Matsumiya G, Iwai S, Ono M, Hata H, Yamauchi T, Nishimura M, Fujino Y, Matsuda H. Effect of a polymorphonuclear elastase inhibitor (sivelestat sodium) on acute lung injury after cardiopulmonary bypass: findings of a double-blind randomized study. Surg Today. 2006;36(4):321-6. doi: 10.1007/s00595-005-3160-y. PMID 16554988
- [Result] Niino T, Hata M, Sezai A, Yoshitake I, Unosawa S, Fujita K, Shimura K, Osaka S, Minami K. Efficacy of neutrophil elastase inhibitor on type A acute aortic dissection. Thorac Cardiovasc Surg. 2010 Apr;58(3):164-8. doi: 10.1055/s-0029-1240846. Epub 2010 Apr 7. PMID 20376727
- [Result] Toyama S, Hatori F, Shimizu A, Takagi T. A neutrophil elastase inhibitor, sivelestat, improved respiratory and cardiac function in pediatric cardiovascular surgery with cardiopulmonary bypass. J Anesth. 2008;22(4):341-6. doi: 10.1007/s00540-008-0645-z. Epub 2008 Nov 15. PMID 19011770
- [Result] Nomura N, Asano M, Saito T, Nakayama T, Mishima A. Sivelestat attenuates lung injury in surgery for congenital heart disease with pulmonary hypertension. Ann Thorac Surg. 2013 Dec;96(6):2184-91. doi: 10.1016/j.athoracsur.2013.07.017. Epub 2013 Sep 25. PMID 24075485
- [Result] Inoue N, Oka N, Kitamura T, Shibata K, Itatani K, Tomoyasu T, Miyaji K. Neutrophil elastase inhibitor sivelestat attenuates perioperative inflammatory response in pediatric heart surgery with cardiopulmonary bypass. Int Heart J. 2013;54(3):149-53. doi: 10.1536/ihj.54.149. PMID 23774238
- [Result] Kohira S, Oka N, Inoue N, Itatani K, Hanayama N, Kitamura T, Fujii M, Takeda A, Oshima H, Tojo K, Yoshitake S, Miyaji K. Effect of the neutrophil elastase inhibitor sivelestat on perioperative inflammatory response after pediatric heart surgery with cardiopulmonary bypass: a prospective randomized study. Artif Organs. 2013 Dec;37(12):1027-33. doi: 10.1111/aor.12103. Epub 2013 Jul 3. PMID 23834653
- [Result] Kohira S, Oka N, Inoue N, Itatani K, Kitamura T, Horai T, Oshima H, Tojo K, Yoshitake S, Miyaji K. Effect of additional preoperative administration of the neutrophil elastase inhibitor sivelestat on perioperative inflammatory response after pediatric heart surgery with cardiopulmonary bypass. Artif Organs. 2014 Dec;38(12):1018-23. doi: 10.1111/aor.12311. Epub 2014 Apr 21. PMID 24750107
- [Result] Fujii M, Miyagi Y, Bessho R, Nitta T, Ochi M, Shimizu K. Effect of a neutrophil elastase inhibitor on acute lung injury after cardiopulmonary bypass. Interact Cardiovasc Thorac Surg. 2010 Jun;10(6):859-62. doi: 10.1510/icvts.2009.225243. Epub 2010 Mar 30. PMID 20354035
- [Result] Abe T, Usui A, Oshima H, Akita T, Ueda Y. A pilot randomized study of the neutrophil elastase inhibitor, Sivelestat, in patients undergoing cardiac surgery. Interact Cardiovasc Thorac Surg. 2009 Aug;9(2):236-40. doi: 10.1510/icvts.2009.206193. Epub 2009 May 15. PMID 19447800
- [Result] Yamashiro S, Arakaki R, Kise Y, Kuniyoshi Y. Prevention of Pulmonary Edema after Minimally Invasive Cardiac Surgery with Mini-Thoracotomy Using Neutrophil Elastase Inhibitor. Ann Thorac Cardiovasc Surg. 2018 Feb 20;24(1):32-39. doi: 10.5761/atcs.oa.17-00102. Epub 2017 Nov 8. PMID 29118307
- [Result] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957